CLINICAL TRIAL: NCT05769439
Title: Hydroxymethylation, Incident Type 2 Diabetes and Incident Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Des Moines University (Other)
Collaborators: Indiana University (Other); Penn State University (Other); EpiGenTek, LLC (Unknown)
Responsible Party: Principal Investigator, Jun Dai, Professor, Des Moines University
Other Study IDs: 1R15HL152330-01A1 (NIH)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Incident Type 2 Diabetes; Incident Obesity
Keywords: hydroxymethylation; twin; monozygotic; dizygotic; fraternal; identical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat DNA samples were collected in the mid-1980. This study used the discordant twin design, a specific nested case-co-twin control design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NTS iT2D-dTwin case-co-twin-control cohort: The twin pairs discordant for incident type 2 diabetes (iT2D) [17 monozygotic (MZ) and 20 dizygotic twin pairs (DZ)] are included from the National Heart, Lung, and Blood Institute (NHLBI) Twin Study (NTS). In a discordant twin pair, one co-twin developed iT2D while his co-twin did not or develop iT2D at least one year later.
  Interventions: Other: No intervention in an observational study
- NTS iOB-dTwin case-co-twin-control cohort: The twin pairs discordant for incident obesity (iOB) [11 monozygotic (MZ) and 15 dizygotic twin pairs (DZ)] are included from the National Heart, Lung, and Blood Institute (NHLBI) Twin Study (NTS). In a discordant twin pair, one co-twin developed iOB while his co-twin did not or develop iOB at least one year later.
  Interventions: Other: No intervention in an observational study

INTERVENTIONS:
Other: No intervention in an observational study — This study is an observational study only.

SUMMARY:
The proposed discordant identical and fraternal twin study of incident type 2 diabetes and incident obesity is pivotal to public health because this study design compares diseased twins with their non-diseased co-twins for a better understanding of environment-induced hydroxymethylation independent of genetic influences as the novel biological mechanism underlying the diseases. By engaging students in the proposed co-twin control study, we will prepare our next generation of public health researchers to sustain our impact on public health across generations. The discovery of new environmentally and epigenetically therapeutic and preventive regimens will pave the way to fight against incident type 2 diabetes and incident obesity.

DETAILED DESCRIPTION:
Hydroxymethylated cytosine (5hmC) in DNA is an epigenetic modification that regulates gene transcription. Type 2 diabetes (T2D) and obesity (OB) are diseases that are serious global public health challenges. Little is known about the role of 5hmC in the development of T2D and OB. In our exploratory study to investigate hydroxymethylation using a co-twin control design, we included three monozygotic twin pairs (MZ) discordant for incident T2D (iT2D) and five separate MZ pairs discordant for prevalent OB from our previous R21 (1R21HL127368-01) study of cardiovascular disease. Using circulating 5hmC as an aggregate surrogate for cumulative systemic hydroxymethylation, intriguingly, we found statistically significant, whole-genome differentially hydroxymethylated regions (DhMRs) related to iT2D and prevalent OB, respectively, after controlling for genetic variation in germline consisting of 3.2 billion base pairs, age-period-cohort effects, and multiple-testing. Due to the very limited sample size and lack of twin pairs discordant for incident OB (iOB) in our prior exploratory study, it is imperative to perform the prospective research in a relatively large sample to generate strong evidence. The National Heart, Lung, and Blood Institute (NHLBI) Twin Study is a well-characterized, 46-year follow-up study initiated in 1969. Leveraging existing rich resources in the NHLBI Twin Study and our established, multi-mechanism students' research engagement plan, we propose this R15 study. Our overall objectives are to characterize circulating 5hmC in relation to iT2D and iOB and to offer an excellent opportunity for students to be engaged in public health epigenome research. These objectives will be achieved by pursuing three specific aims: 1) measure whole genome hydroxymethylation (5hmC) in blood DNA samples; 2) test if DNA regions are differentially hydroxymethylated in relation to iT2D (aim 2-1) and iOB (aim 2-2) independent of germline and common environment; which, in turn, will identify novel differentially hydroxymethylated regions; and 3) characterize sociobehavioral and other environmental correlates of hydroxymethylation in literature-based candidate and novel DNA regions independent of germline and common environment. We will include all available twin pairs discordant for iT2D [17 MZ and 20 dizygotic twin pairs (DZ)] and separate twin pairs discordant for iOB (11 MZ pairs and 15 DZ pairs) from NHLBI Twin Study. The NHLBI Twin Study twins were born between 1917 and 1927, a period when 2 male MZ pairs and 4 male DZ pairs of twins were born per 1,000 live births. An illustrative example is that inclusion of our dMZ twin sample size is equivalent to that of at least 126,746 singletons. The significance of our study is to provide innovative evidence about iT2D and iOB-discriminating hydroxymethylation induced environmentally, which could impact disease prevention and treatment through the improvement of modifiable environmental factors. Our study will offer a unique opportunity for engaging medical and graduate students at the applicant's institute in the public health epigenome research.

ELIGIBILITY:
Inclusion Criteria:

In the NHLBI Twin Study, middle-aged, male, veteran twins were recruited at baseline (1969-1973).

Inclusion criteria include 1) an iT2D-discordant MZ and DZ twin pair in which one co-twin subsequently became diabetic after exam 3 through December 31, 2015 (i.e., case twin) while the other co-twin was nondiabetic on the index date (i.e., control twin); 2) an iOB-discordant MZ and DZ twin pair in which both co-twins were non-obese at exam 3 and one co-twin subsequently became obese55 after exam 3 through exam 5 (i.e., case twin) while the other co-twin was non-obese on the index date (i.e., control twin); 3) all twins must have blood DNA samples available and collected at least one year prior to the index date for each of the specific diseases (i.e., iT2D and iOB); and participant's date of birth, vital status, cause of death, death date, and date for the blood DNA collection are available.

Exclusion Criteria:

-

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Below is the Parent Cohort Description:
  The NHLBI Twin Study (NTS) is a prospective study of the genetic and environmental etiology of cardiovascular disease. Initiated in 1969, researchers recruited 514 white male twin pairs (i.e., 1,024 men) born between 1917 and 1927. The twins were roughly 50% monozygotic twin pairs (MZ) and 50% dizygotic twin pairs (DZ) and were middle-aged at baseline (1969-1973). The five research sites were Framingham, MA; San Francisco, CA; Davis, CA; Los Angeles, CA; and Indianapolis, IN. The participant inclusion criterion was the geographic proximity to the study sites (within 100 miles in New England and California, and within 200 miles of Indianapolis, Indiana). The twins received physical examinations based on the renowned Framingham Heart Study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
novel differentially hydroxymethylated regions (DhMRs) concerning incident type 2 diabetes | April 1, 2023 to December 31, 2023
  Whole-genome 5hmC will be measured among MZ and DZ twin pairs discordant for incident type 2 diabetes
novel DhMRs concerning incident obesity | April 1, 2023 to December 31, 2023
  Whole-genome 5hmC will be measured among MZ and DZ twin pairs discordant for incident obesity
evidence-based DhMRs concerning incident type 2 diabetes | May1, 2022 to December 31, 2023
  literature review will be performed to find the candidate DhMRs
evidence-based DhMRs concerning incident obesity | May1, 2022 to December 31, 2023
  literature review will be performed to find the candidate DhMRs

CONTACTS AND LOCATIONS:
Overall Officials: Jun Dai, MD, PhD, Principal Investigator — Des Moines University
Locations (1):
- Des Moines University, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Data Sharing Plan:
  All investigators will adhere to the NIH policies for data sharing. De-identified data will be available and shared commonly 6 months after the investigators' quality manuscript is accepted. The data sharing agreement will be required. We will also share data through presentations at scientific meetings, research seminars, and publications of manuscripts.
  Genomic Data Sharing Plan (GDS) This application generates whole genome hydroxymethylation using the enrichment-based method followed by NextGen-seq. These data will be shared with investigators who prepare a manuscript.